CLINICAL TRIAL: NCT07272681
Title: Effect of Helicobacter Pylori Eradication on Gastrointestinal Symptoms in Adult Patients
Brief Title: Effect of H. Pylori Eradication on The Improvement of Gastrointestinal Symptoms
Acronym: HPE-GI
Status: Not yet recruiting | Type: Observational
Sponsor: Amany Usama Ahmed Arafa (Other)
Responsible Party: Sponsor-Investigator, Amany Usama Ahmed Arafa, Resident doctor, Tropical Medicine and Gastroenterology, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med--25-11-1MS
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Helicobacter Pylori Infection; Dyspepsia; Gastrointestinal Symptoms
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- H. pylori-positive adults - Eradication therapy group - Adult patients with H. pylori infection: Adult patients with confirmed Helicobacter pylori infection who have received standard eradication therapy prescribed by their healthcare providers. The study will observe and evaluate changes in gastrointestinal symptoms after completion of the prescribed treatment, without altering or influencing the treatment regimen.

SUMMARY:
This study aims to evaluate the effect of Helicobacter pylori eradication on gastrointestinal symptoms in adult patients. H. pylori infection is a common cause of dyspepsia and other upper gastrointestinal complaints. The trial will assess whether successful eradication therapy leads to significant improvement in symptoms compared to baseline. Adult patients diagnosed with H. pylori infection will receive standard eradication treatment, and symptom changes will be monitored using validated questionnaires over a defined follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older.
2. Confirmed diagnosis of Helicobacter pylori infection by one or more diagnostic tests.
3. Presence of any upper or lower gastrointestinal symptoms.
4. Willingness to undergo H. Pylori eradication therapy and follow-up.
5. Ability to provide informed consent.

Exclusion Criteria:

1. Age less than 18 years.
2. The previously unsuccessful application of empirical H. pylori eradication therapy.
3. Use of non-steroidal anti-inflammatory drugs (NSAIDs).
4. Any malignant disease of the stomach or any other site.
5. Any associated comorbidity (renal insufficiency, mental illness).
6. History of allergies to proton pump inhibitors or antibiotics.
7. Refusal to participate in the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult patients (≥18 years) diagnosed with Helicobacter pylori infection by invasive or non-invasive tests (urea breath test or stool antigen test) and who have completed standard eradication therapy prescribed by their healthcare providers. The population includes both male and female patients presenting with gastrointestinal symptoms such as dyspepsia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in gastrointestinal symptoms after Helicobacter pylori eradication. | 6 weeks
  Gastrointestinal symptom improvement will be assessed using the Gastrointestinal Symptom Rating Scale (GSRS).
  The GSRS consists of 15 items, each scored from 1 to 7, giving a total score range of:
  Minimum score: 1 (absence of symptoms) Maximum score: 7 (most severe symptoms) Higher scores indicate worse gastrointestinal symptoms. Change will be calculated by comparing baseline scores to follow-up scores after completion of eradication therapy.
Eradication success rate. | 8 weeks
  Proportion of patients achieving confirmed eradication of Helicobacter pylori using non-invasive testing (either urea breath test or stool antigen test), performed after completing eradication therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Amany Usama, Principal Investigator — Department of Gastroenterology and Tropical medicine Sohag University Hospital

IPD SHARING:
Plan to Share IPD: Undecided